CLINICAL TRIAL: NCT06098573
Title: Development and Evaluation of 'High Alert', a Mobile-Based Brief Intervention to Reduce Driving Under the Influence of Cannabis Among Youth
Brief Title: Development and Evaluation of HighAlert
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123368
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cannabis; Youth Drinking
MeSH Terms: conditions — Marijuana Abuse; Underage Drinking | interventions — Medication Errors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Program 1: High Alert (Experimental): High Alert
  Interventions: Behavioral: High Alert
- Program 2: Information condition (Active Comparator): Active Control- Information condition
  Interventions: Behavioral: Information condition
- No contact (Placebo Comparator): Passive control- No contact
  Interventions: Behavioral: No contact

INTERVENTIONS:
Behavioral: High Alert — Participants assigned to the 'High Alert' condition will complete four interactive modules using their smartphones. These modules are hosted online via the Computerized Intervention Authoring Software, version 3.0 (https://www.cias.app [CIAS]). CIAS is a non- commercial, easily modifiable, web-based intervention platform used widely in the digital substance use literature. No identifiable information is requested or stored in CIAS. This program is only intended to deliver the content interactively. None of the questions asked in CIAS will be treated as research data. We will only report on the proportion of questions answered by participants (as a measure of adherence). Individual responses to questions will not be analyzed nor reported on. The purpose of the questions is for participants to engage with the content interactively
  Arms: Program 1: High Alert
Behavioral: Information condition — Participants in the DUIC Information condition will receive a Qualtrics link with six infographics created to educate about DUIC. Four infographics were retrieved from government websites, one was provided by a non-profit (i.e., Arrive Alive Drive Sober), and the research team created the final one. After reviewing each infographic, participants will respond to a few questions about the infographic. Questions asked to the DUIC Info Control will obtain data related to: seeing the infographic before, perceptions on the infographic content, aspects they liked/disliked, and likelihood to share with their peers. All items will be treated as research data.
  Arms: Program 2: Information condition
Behavioral: No contact — Participants in the passive control will receive no contact until the three and six-month follow-ups.
  Arms: No contact

SUMMARY:
In Canada, youth ages 16-24 have the highest rates of cannabis use, impaired driving, and express the least concern for driving under the influence of cannabis (DUIC). As such, developing effective and practical DUIC prevention efforts is crucial. This study aims to evaluate the effects of 'High Alert' in reducing 3-month risky cannabis use and DUIC among young Ontarian drivers. 'High Alert' is an interactive web-based smartphone application developed by the research team with the feedback of experts and youth. 'High Alert' modules focus on recognizing what constitutes risky cannabis use, the effects of cannabis on driving, the risks of DUIC, and strategies to avoid DUIC. A pilot randomized controlled trial will compare the effects of 'High Alert' with an active control (DUIC Information) and passive control (no contact). Overall, effectively preventing DUIC among youth is critically needed and time-sensitive.

ELIGIBILITY:
Inclusion:

* ages 18-24
* valid Ontario driver's license
* access to a motor vehicle
* report DUIC at least three times in the past three months
* proficient in English
* have a smartphone they can complete the intervention with.

Exclusion Criteria:

* Individuals under 18 and those over 24
* resides outside Ontario
* non-drivers

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Past driving under the influence of cannabis | 3-months
  "in the past three months, how many times have you driven within two hours of inhaling cannabis or within four hours of ingesting cannabis". Continuous variable (min=0, no maximum). Higher numbers indicate worse outcome (i.e., more impaired driving).

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No